CLINICAL TRIAL: NCT01101061
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 785 in Healthy Postmenopausal Japanese Women
Brief Title: A Single-dose Study Evaluating Romosozumab (AMG 785) in Healthy Postmenopausal Japanese and Non-Japanese Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20090378
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Osteopenia
Keywords: Amgen; Phase 1; Postmenopausal; Japanese
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Romosozumab (Experimental): Japanese women in cohorts 1, 2, and 4 will receive a single dose of 1, 3, or 5 mg/kg romosozumab. Non-Japanese women in cohort 3 will receive a single dose of 3 mg/kg romosozumab.
  Interventions: Drug: Romosozumab
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Romosozumab — Administered by subcutaneous injection
  Other Names: AMG 785; EVENITY™
  Arms: Romosozumab
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the safety, tolerability and potential immune response to romosozumab following single subcutaneous (SC; injection under the skin) dose administration in healthy postmenopausal Japanese and non-Japanese women.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects must be first (4 grandparents, biologic parents and subject born in Japan), second (4 grandparents and biological parents born in Japan) or third (4 grandparents born in Japan) generation Japanese
* Body mass index ≤ 25 kg/m², inclusive at screening
* Postmenopausal females defined as 12 continuous months of spontaneous amenorrhea confirmed by a serum follicle-stimulating hormone (FSH) result > 40 mIU/mL, or 6 weeks postsurgical bilateral oophorectomy (with or without hysterectomy) as documented in medical history (verified with an operative note, if available)

Exclusion Criteria:

* Osteoporosis, as defined by bone mineral density (BMD) T-scores of the lumbar spine (L1-L4) or total evaluable vertebrae (if fewer than L1-L4); or femoral neck ≤ -2.5
* History of vertebral fracture or fragility fracture of the wrist, humerus, hip or pelvis;
* Diagnosed with any condition that will affect bone metabolism

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-05-03 (Actual); Primary Completion 2010-11-01 (Actual); Study Completion 2010-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 study centers in the United States. Eligible participants were healthy, postmenopausal first, second, or third generation Japanese women and non-Japanese women residing in the United States.
Pre-assignment Details: Participants were assigned to one of 4 cohorts. In 3 of the cohorts Japanese women were randomized in a 3:1 ratio to receive 1, 3, or 5 mg/kg romosozumab or placebo. In a 4th cohort non-Japanese women were randomized in a 2:1 ratio to receive 3 mg/kg romosozumab or placebo.
Groups:
- Japanese Women: Placebo: Japanese participants received a single subcutaneous injection of placebo on day 1.
- Japanese Women: Romosozumab 1 mg/kg: Japanese participants received a single subcutaneous injection of 1 mg/kg romosozumab on day 1.
- Japanese Women: Romosozumab 3 mg/kg: Japanese participants received a single subcutaneous injection of 3 mg/kg romosozumab on day 1.
- Japanese Women: Romosozumab 5 mg/kg: Japanese participants received a single subcutaneous injection of 5 mg/kg romosozumab on day 1.
- Non-Japanese Women: Placebo: Non-Japanese participants received a single subcutaneous injection of placebo on day 1.
- Non-Japanese Women: Romosozumab 3 mg/kg: Non-Japanese participants received a single subcutaneous injection of 3 mg/kg romosozumab on day 1.
Period: Overall Study
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
Started | 6 | 6 | 7 | 6 | 2 | 4
Received Study Drug | 6 | 6 | 6 | 6 | 2 | 4
Completed | 6 | 6 | 6 | 6 | 2 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 4 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 6 | 3 | 2 | 4 | 24
  >=65 years | 2 | 1 | 0 | 3 | 0 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (5.7) | 59.3 (4.9) | 61.7 (3.0) | 59.7 (7.7) | 57.5 (3.5) | 55.0 (4.8) | 59.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 6 | 2 | 4 | 30
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6 | 6 | 6 | 6 | 1 | 0 | 25
  White | 0 | 0 | 0 | 0 | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: A serious adverse event (SAE) is defined as an adverse event that
  * is fatal
  * is life threatening
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * other significant medical hazard. A treatment-related AE is any treatment-emergent AE that per investigator review has a reasonable possibility of being caused by the investigational product.
Time Frame: Participants who received a 1 or 3 mg/kg dose (romosozumab or placebo) were followed for 2 months (day 57) after study drug administration and participants who received 5 mg/kg were followed for 3 months (day 85) for safety assessments.
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 4
Participants
  Any adverse event | 6 | 4 | 3 | 6 | 2 | 4
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse events | 2 | 1 | 2 | 1 | 0 | 0
  AEs leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Developed Anti-romosozumab Binding Antibodies
Description: Participants who were negative for anti-romosozumab binding antibodies at baseline with a positive result at any time post-baseline.
Time Frame: Day 29, and end of study (day 57 for participants assigned to 1 or 3 mg/kg romosozumab/placebo or day 85 for participants assigned to 5 mg/kg romosozumab/placebo)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Serum Calcium Levels
Time Frame: Baseline, days 2, 3, 4, 6, 8, 12, 22, 29, 43, 57, 71, and 85
Population: All treated participants; only participants in the 5 mg/kg cohort were assessed at days 71 and 85.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 4
mmol/L
  Baseline | 2.34 (0.04) | 2.31 (0.04) | 2.33 (0.03) | 2.38 (0.03) | 2.28 (0.08) | 2.45 (0.04)
  Day 2 | 2.33 (0.04) | 2.34 (0.03) | 2.31 (0.03) | 2.36 (0.03) | 2.34 (0.04) | 2.40 (0.05)
  Day 3 | 2.33 (0.05) | 2.36 (0.04) | 2.31 (0.03) | 2.38 (0.03) | 2.34 (0.01) | 2.43 (0.03)
  Day 4 | 2.32 (0.05) | 2.31 (0.03) | 2.30 (0.03) | 2.32 (0.03) | 2.38 (0.02) | 2.36 (0.04)
  Day 6 | 2.39 (0.05) | 2.30 (0.03) | 2.31 (0.04) | 2.35 (0.04) | 2.28 (0.02) | 2.40 (0.03)
  Day 8 | 2.39 (0.05) | 2.25 (0.02) | 2.31 (0.03) | 2.29 (0.03) | 2.35 (0.00) | 2.38 (0.03)
  Day 12 | 2.35 (0.06) | 2.27 (0.05) | 2.33 (0.03) | 2.28 (0.02) | 2.33 (0.03) | 2.28 (0.04)
  Day 22 | 2.31 (0.03) | 2.31 (0.03) | 2.28 (0.05) | 2.25 (0.03) | 2.33 (0.00) | 2.36 (0.03)
  Day 29 | 2.37 (0.03) | 2.30 (0.04) | 2.28 (0.03) | 2.30 (0.02) | 2.36 (0.04) | 2.38 (0.05)
  Day 43 | 2.35 (0.04) | 2.33 (0.03) | 2.28 (0.03) | 2.34 (0.04) | 2.30 (0.07) | 2.34 (0.01)
  Day 57 | 2.37 (0.03) | 2.32 (0.04) | 2.29 (0.04) | 2.30 (0.03) | 2.28 (0.00) | 2.31 (0.02)
  Day 71: number analyzed (Participants) | 6 | 0 | 0 | 6 | 0 | 0
  Day 71 | 2.34 (0.01) |  |  | 2.39 (0.02) |  |
  Day 85: number analyzed (Participants) | 2 | 0 | 0 | 6 | 0 | 0
  Day 85 | 2.29 (0.01) |  |  | 2.35 (0.02) |  |

4. Primary Outcome: Serum Intact Parathyroid Hormone (iPTH) Levels
Time Frame: Baseline and days 2, 3, 4, 6, 8, 12, 22, 29, 43, 57, 71, and 85
Population: All treated participants; only participants in the 5 mg/kg cohort were assessed at days 71 and 85
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 4
pmol/L
  Baseline | 4.47 (0.97) | 4.24 (0.70) | 4.93 (0.84) | 3.63 (0.62) | 3.77 (1.65) | 2.73 (0.37)
  Day 2 | 4.51 (0.78) | 4.92 (0.78) | 5.01 (0.47) | 4.23 (0.54) | 3.50 (1.49) | 2.57 (0.23)
  Day 3 | 4.93 (0.71) | 4.69 (0.69) | 5.38 (0.44) | 4.58 (0.76) | 3.50 (1.06) | 2.89 (0.37)
  Day 4 | 4.47 (0.84) | 5.09 (0.69) | 5.09 (0.23) | 5.20 (1.13) | 3.93 (1.70) | 3.55 (0.73)
  Day 6 | 4.21 (0.67) | 4.97 (0.93) | 5.75 (0.72) | 4.44 (0.77) | 3.82 (1.49) | 3.66 (0.66)
  Day 8 | 4.19 (0.95) | 5.91 (0.86) | 5.23 (0.68) | 4.79 (0.90) | 4.14 (1.91) | 3.98 (0.68)
  Day 12 | 5.04 (0.95) | 6.42 (0.59) | 5.46 (0.41) | 5.80 (0.61) | 4.19 (1.86) | 4.46 (0.64)
  Day 22 | 4.69 (0.74) | 5.57 (0.64) | 6.15 (0.56) | 7.09 (0.84) | 5.46 (2.71) | 4.62 (0.68)
  Day 29 | 4.83 (0.99) | 5.02 (0.74) | 5.92 (0.68) | 6.14 (0.72) | 4.83 (2.81) | 4.43 (0.40)
  Day 43 | 4.61 (0.89) | 6.03 (0.73) | 5.27 (0.32) | 5.61 (0.84) | 3.93 (1.27) | 3.53 (0.35)
  Day 57 | 3.89 (0.84) | 4.90 (0.64) | 4.87 (0.39) | 4.86 (0.55) | 2.76 (0.85) | 2.68 (0.27)
  Day 71: number analyzed (Participants) | 6 | 0 | 0 | 6 | 0 | 0
  Day 71 | 3.40 (0.85) |  |  | 4.10 (0.47) |  |
  Day 85: number analyzed (Participants) | 2 | 0 | 0 | 6 | 0 | 0
  Day 85 | 3.02 (0.80) |  |  | 3.82 (0.58) |  |

5. Secondary Outcome: Maximum Percent Change From Baseline in Serum Procollagen Type 1 N-terminal Propeptide (P1NP)
Time Frame: Baseline and days 2, 3, 4, 6, 8, 12, 22, 29, 43, 57, 71, and 85
Population: All treated participants
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 4
percent change | 26.85 (6.39) | 59.23 (12.21) | 102.57 (18.26) | 196.37 (29.79) | 8.30 (1.78) | 164.44 (35.58)

6. Secondary Outcome: Maximum Percent Change From Baseline in Serum C-telopeptide (CTX)
Time Frame: Baseline and days 2, 3, 4, 6, 8, 12, 22, 29, 43, 57, 71, and 85
Population: All treated participants
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 4
percent change | -12.64 (1.40) | -16.19 (7.36) | -35.92 (1.94) | -39.17 (5.13) | -25.46 (8.52) | -43.32 (9.96)

7. Secondary Outcome: Percent Change From Baseline in Sclerostin
Time Frame: Baseline and days 12, 29, 43, 57, 71, and 85
Population: All treated participants; only participants in the 5 mg/kg cohort were assessed at days 71 and 85.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 2 | 4
percent change
  Day 12 | -3.78 (3.72) | 6639.01 (534.50) | 13749.61 (1091.63) | 17028.81 (1875.81) | -17.95 (6.38) | 14652.96 (1349.38)
  Day 29 | 591.80 (596.47) | 1602.70 (231.77) | 7667.80 (675.45) | 12723.54 (2138.65) | -14.54 (1.78) | 9581.13 (1283.73)
  Day 43 | -15.43 (11.39) | 467.07 (55.62) | 3384.02 (613.99) | 6844.74 (1730.04) | -9.35 (4.59) | 4487.33 (1771.30)
  Day 57 | -17.89 (11.96) | 167.37 (28.33) | 911.23 (156.09) | 2836.61 (1109.97) | -0.41 (12.65) | 1826.83 (917.98)
  Day 71: number analyzed (Participants) | 2 | 0 | 0 | 6 | 0 | 0
  Day 71 | -39.80 (3.87) |  |  | 997.02 (532.06) |  |
  Day 85: number analyzed (Participants) | 2 | 0 | 0 | 6 | 0 | 0
  Day 85 | -27.41 (2.02) |  |  | 415.38 (243.40) |  |

8. Secondary Outcome: Time to Maximum Observed Concentration of Romosozumab
Description: Serum concentrations of romosozumab were measured using a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) was 50 ng/mL.
Time Frame: Predose, 12 hours postdose, and on days 2, 3, 4, 6, 8, 12, 22, 29, 43, and 57, and days 71 and 85 for participants assigned tp 5 mg/kg romosozumab/placebo.
Population: All treated participants who received romosozumab
Measure: Median (Full Range); unit: days
Arm/Group | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 4
days | 5.0 [5.0 to 8.0] | 5.0 [3.0 to 12] | 5.0 [5.0 to 7.0] | 5.0 [5.0 to 7.0]

9. Secondary Outcome: Maximum Observed Concentration of Romosozumab
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All treated participants who received romosozumab
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 4
µg/mL | 4.06 (1.45) | 17.1 (4.7) | 33.8 (8.1) | 18.6 (1.1)

10. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUClast) of Romosozumab
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All treated participants who received romosozumab
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 4
µg*day/mL | 64.0 (27.0) | 344 (90) | 804 (320) | 412 (136)

11. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUCinf) for Romosozumab
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All treated participants who received romosozumab
Measure: Mean (Standard Deviation); unit: µg*day/mL
Arm/Group | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 4
µg*day/mL | 64.7 (26.8) | 347 (90) | 806 (323) | 421 (147)

12. Secondary Outcome: Apparent Clearance (CL/F) of Romosozumab
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All treated participants who received romosozumab
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 4
mL/day/kg | 18.6 (10.0) | 9.27 (2.64) | 6.98 (2.35) | 7.91 (2.68)

13. Secondary Outcome: Half-life Associated With Beta (Plateau) Phase of Elimination (T1/2,β) for Romosozumab
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All treated participants who received romosozumab with available T1/2,β data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 0 | 1 | 6 | 2
days |  | 15.1 (NA) — Could not be calculated for 1 participant | 16.2 (4.1) | 15.3 (6.2)

14. Secondary Outcome: Half-life Associated With Gamma (Terminal) Phase of Elimination (T1/2,ɣ) for Romosozumab
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All treated participants who received romosozumab
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Romosozumab 3 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 4
days | 5.82 (1.05) | 6.31 (1.14) | 7.19 (1.55) | 6.81 (2.69)

ADVERSE EVENTS:
Time Frame: Participants who received a 1 or 3 mg/kg dose (romosozumab or placebo) were followed for 2 months (day 57) after study drug administration and participants who received 5 mg/kg were followed for 3 months (day 85) for safety assessments
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Japanese Women: Placebo | Japanese Women: Romosozumab 1 mg/kg | Japanese Women: Romosozumab 3 mg/kg | Japanese Women: Romosozumab 5 mg/kg | Non-Japanese Women: Placebo | Non-Japanese Women: Romosozumab 3 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/6 | 3/6 | 6/6 | 2/2 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Japanese Women: Placebo (N=6) | Japanese Women: Romosozumab 1 mg/kg (N=6) | Japanese Women: Romosozumab 3 mg/kg (N=6) | Japanese Women: Romosozumab 5 mg/kg (N=6) | Non-Japanese Women: Placebo (N=2) | Non-Japanese Women: Romosozumab 3 mg/kg (N=4)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 2 | 1 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 2 | 1 | 1 | 1 | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Venomous sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 3 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.